CLINICAL TRIAL: NCT01492959
Title: A Prospective, Open, Uncontrolled, Observational Study With Innolet in Daily Clinical Situations According to the Product Labelling, Without Any Study Specific Investigations
Brief Title: Observational Study With InnoLet® in Daily Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INNOLET-1888
Record Dates: First submitted 2011-12-09; First posted 2011-12-15 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin human
  Interventions: Drug: insulin human

INTERVENTIONS:
Drug: insulin human — Insulin human delivered with the InnoLet® device was prescribed according to product labelling to subjects in need of insulin treatment

SUMMARY:
This study is conducted in Asia. The aim of this study is to review the efficacy and safety of insulin treatment with InnoLet® in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (Type 1 or type 2)
* Need insulin treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean patients with diabetes mellitus in need of insulin treatment
Sampling Method: Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2004-03-23 (Actual); Primary Completion 2005-03-23 (Actual); Study Completion 2005-03-23 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Adverse events: Serious and non-serious

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com